CLINICAL TRIAL: NCT04623918
Title: Randomized Trial of Iron-Biofortified Rice in Women in the Philippines
Brief Title: Iron-Biofortified Rice Intervention in the Philippines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: Penn State University (Other); University of the Philippines (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Haas2005
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Iron-deficiency; Anemia
Keywords: Anemia; Iron; Biofortification; Philippines; Iron deficiency; Women of reproductive age
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia; Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masking description: The study was a double-blind, randomized controlled trial of; (1) iron-biofortified rice (IR68144-2B-2-2-3), compared to (2) a commercially available variety of rice (C4), with the intervention randomized at the individual level. Administrators, participants, research staff (i.e. responsible for daily data collection and preparation of rice for all meals, assessment of outcomes), and laboratory staff were blinded to the intervention group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron-biofortified rice (Experimental): Iron-biofortified rice (IR68144-2B-2-2-3)
  Interventions: Other: Iron-biofortified rice
- Control rice (Active Comparator): Control rice (C4)
  Interventions: Other: Control rice

INTERVENTIONS:
Other: Iron-biofortified rice — Iron-biofortified rice (IR68144-2B-2-2-3)
  Arms: Iron-biofortified rice
Other: Control rice — Control rice (C4), identical in appearance
  Arms: Control rice

SUMMARY:
The objective of this randomized efficacy feeding trial was to determine the effects of consuming iron-biofortified rice on iron status in women, compared to non-biofortified rice. A randomized trial of biofortified rice (IR68144-2B-2-2-3), bred to enhance iron content, was conducted among women living in convents in the greater area of Manila, Philippines for 9 months.

DETAILED DESCRIPTION:
Iron deficiency is the most prevalent nutritional deficiency globally, with the highest burden in women of reproductive age and children. In this randomized controlled trial, 317 women aged 18-45 years living in convents in the greater Manila area, Philippines, were fed meals using either biofortified or commercially available rice for all meals, 7 days a week, for 9 months. Women living in convents in the greater Manila area were recruited for this study. These women represent a segment of the population at high risk for iron deficiency, consume large quantities of rice, and all of their meals are prepared and consumed in common kitchen and dining areas, respectively.

The investigators hypothesized that daily consumption of iron-biofortified rice (IR68144-2B-2-2-3) would improve hemoglobin, serum ferritin, and total body iron in 9 months, compared to control rice. In order to examine this hypothesis, the investigators conducted a randomized efficacy trial of iron-biofortified rice and iron status in among women living in convents in the greater area of Manila, Philippines for 9 months.

The objective of this randomized efficacy feeding trial was to determine the effects of consuming iron-biofortified rice on iron status in women, compared to non-biofortified rice.

The long-term goal of this study is to determine if iron bio-fortification of rice is an efficacious and potentially effective strategy to improve iron status of at-risk populations in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* Women (18-45 years old) living in convents in the greater Manila area
* Hb ≥10.5 g/dL

Exclusion Criteria:

* Current or history of gastrointestinal or hematological disorders
* Taking iron supplements or medications that could interfere with hematopoiesis or dietary iron absorption
* Hb <10.5 g/dL
* Women expressed uncertainty in their ability to participate for the full (9 month) trial

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 288 (Actual)
Dates: Start 2002-06-01 (Actual); Primary Completion 2003-12-31 (Actual); Study Completion 2003-12-31 (Actual)

PRIMARY OUTCOMES:
Change in serum ferritin | 9 months
  Serum ferritin (SF)
Change in sTfR | 9 months
  Soluble transferrin receptor (sTfR)
Change in TBI | 9 months
  Total body iron (TBI)

SECONDARY OUTCOMES:
Change in hemoglobin among women who were anemic at baseline | 9 months
  Changes in hemoglobin (Hb) in women who were anemic at baseline
Changes in SF among women who were non-anemic at baseline | 9 months
  Changes in SF among women who were non-anemic at baseline
Changes in sTfR among women who were non-anemic at baseline | 9 months
  Changes in sTfR among women who were non-anemic at baseline
Changes in TBI among women who were non-anemic at baseline | 9 months
  Changes in TBI among women who were non-anemic at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jere Haas, Principal Investigator — Cornell University
Locations (1):
- University of the Philippines, Los Baños, Laguna, Philippines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haas JD, Beard JL, Murray-Kolb LE, del Mundo AM, Felix A, Gregorio GB. Iron-biofortified rice improves the iron stores of nonanemic Filipino women. J Nutr. 2005 Dec;135(12):2823-30. doi: 10.1093/jn/135.12.2823. PMID 16317127